CLINICAL TRIAL: NCT04887896
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Assessing the Effect of GS500 in Subjects With Functional Constipation
Brief Title: Assessing GS500 in Functional Constipation
Acronym: TRANSIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gelesis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-500-001
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Constipation - Functional

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, placebo-controlled, parallel-group, flexible-dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GS500 flexible dose (Experimental): 3, 2, or 4 GS500 capsules 2 times per day
  Interventions: Device: GS500
- Placebo flexible dose (Placebo Comparator): 3, 2, or 4 placebo capsules 2 times per day
  Interventions: Device: Placebo

INTERVENTIONS:
Device: GS500 — Device: GS500
  Arms: GS500 flexible dose
Device: Placebo — Device: Placebo
  Arms: Placebo flexible dose

SUMMARY:
This study is designed to evaluate the safety, tolerability and efficacy of GS500 as a superabsorbent hydrogel for relief of constipation in subjects with functional constipation.

DETAILED DESCRIPTION:
To evaluate the safety, tolerabilityand efficacy of GS500 as a superabsorbent hydrogel for relief of constipation in subjects with functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years old
* BMI ≥18.5 and <35 kg/m2
* Rome IV criteria for FC
* Compliant with reporting during Baseline Run-in .
* Ability to record daily bowel habits, including frequency, stool consistency, straining, completeness of evacuation, and patient reported outcomes
* Ability to follow verbal and written instructions
* Consent obtained via signed ICF

Exclusion Criteria:

* Meeting Rome IV criteria for IBSat screening
* Missing > 2 days of daily bowel habits reporting during either week of the Baseline Run-in period
* Patients reporting laxative, enema, and/or suppository usage for >2 days or any usage of a prohibited medication during the Baseline Run-in
* Patients reporting watery stools for any SBM or loose stools for >1 SBM in the absence of laxatives during Baseline Run-in
* Need for routine manual maneuvers in the last 6 months in order to achieve a BM
* History of significant GI lumen surgery at any time or other GI or abdominal surgery except cholecystectomy or appendectomy within 2 months prior to screening
* Documented GI obstruction
* History of laxative abuseas judged by investigator team
* Glycosylated hemoglobin (HbA1c) ≥8.5%
* Known history of Crohn's disease or ulcerative colitis
* Pregnancy in females of childbearing potential or lactation
* Absence of medically approved contraception in females of childbearing potential
* History of allergic reaction to carboxymethylcellulose, citric acid, sodium stearyl fumarate, HPMC, pectin, gelatin, maltotextrin or titanium dioxide
* Currently enrolled in another investigational device or drug study, or less than 3 months since ending another investigational device or drug study(s), or receiving other investigational treatment(s).
* Subjects anticipating surgical intervention during the study
* Angina, coronary bypass, or myocardial infarction within 6 months prior to Screening Visit
* History of swallowing disorders
* History of gastroparesis
* History of intestinal stricture (e.g., Crohn's disease)
* History of intestinal obstruction or subjects at high risk of intestinal obstruction including suspected small bowel adhesions
* History of maltodextrin intolerance
* Presence of metastatic cancer or current use of systemic anti-cancer treatments
* Anticipated requirement for use of prohibited concomitant medications
* Current use of prescribed or illicit opioids
* Use of intestinal secretagogues to treat constipation/IBS within 12 months of the screening visit
* Any other clinically significant disease or biochemical abnormality interfering with the assessments of GS500, according to the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 8 weeks
  Proportion of CSBM Responders defined as subjects with increase of ≥ 1 CSBM from Baseline Run-In during at least 6 of the 8 weeks of the Effectiveness period

SECONDARY OUTCOMES:
Straining score (EoPS) | 8 weeks
Constipation severity (self-assessment on 0 to 10 numerical rating scale) | 8 weeks
SBM stool consistency (BSFS) | 8 weeks
SBM frequency rate (SBMs/week) | 8 weeks
CSBM frequency rate (CSBMs/week) | 8 weeks
Proportion of subjects with increase of ≥2 CSBMduringat least6 of the 8 weeks of the Effectiveness period | 8 weeks

IPD SHARING:
Plan to Share IPD: No